CLINICAL TRIAL: NCT02890511
Title: A Study of DHP107, a Novel Oral Paclitaxel Formulation, to Determine Maximum Tolerated Dose and Recommended Dose for Phase II Trial in Patients With Advanced Solid Cancer
Brief Title: A Study DHP107, a Novel Oral Paclitaxel Formulation, in Patients With Advanced Solid Tumours or Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daehwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107CS-2
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Solid Tumor; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DHP107(Oral paclitaxel) (Experimental): * Phase I (determining MTD) The patients diagnosed with either advanced or metastatic solid cancers were enrolled. The administered dose was escalated in a step-wise manner by an increment of 2 x 50 mg/m2 at each dose level. Three patients were treated for toxicity evaluation for each dose level.
  * Phase IIa (efficacy evaluation) The safety and efficacy of the corresponding dose was investigated more closely by increasing the patient number to 6 or more patients in the dose tentatively determined as recommended dose for phase IIa clinical trial.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Oral administration on day 1,8,15 of 4-week cycle until progression, unacceptable toxicity or withdrawal of informed consent.
  Other Names: DHP107

SUMMARY:
A study of DHP107, a novel oral paclitaxel formulation, to determine maximum tolerated dose and recommended dose for phase II trial in patients with advanced solid cancer and explore efficacy of DHP107 in patients with gastric cancer

DETAILED DESCRIPTION:
1. Primary objective To determine the maximum tolerated dose and the recommended dose for phase 2 clinical trial for the repeated administration of DHP107 (oral paclitaxel) on advanced solid cancer patients
2. Secondary objectives

   * To identify the dose limiting toxicity and the safety (toxicity) of DHP107
   * To evaluate the efficacy (tumor response rate) of DHP107
   * To assess pharmacokinetic (PK) characteristics of DHP107

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 70 years old
2. Patients prognosed with advanced or metastatic solid cancer by histopathology or cytology analysis who have no available standard therapy or who have failed at least once with the standard therapy
3. Adequate bone marrow function, liver function and adequate kidney function
4. Eastern Cooperative Oncology Group performance status ≤ 2
5. Life expectancy of 3 month or more
6. Written informed consent

Exclusion Criteria:

1. Major infectious or neurological disease and bowel obstruction
2. Brain metastasis or hematologic malignancy
3. Patients who underwent surgery, radiation therapy, hormone or chemotherapy within 4 weeks prior to the beginning of investigational drug administration
4. Patients with the history of failure to the taxane line of chemotherapy (with the exception of when it was used before 6 month as adjuvant therapy or when the treatment was discontinued due to docetaxel related side effect)
5. Patients who are required to continuously take P-gp (P-glycoprotein) suppressor, immune suppressor, proton-pump inhibitor or H2-receptor antagonist during clinical trial period
6. Patients deemed by the investigator to suffer from severe heart disease (myocardial infarction, congestive heart failure, arrythmia accompanying drastic changes on ECG, severe or unstable angina pectoris, or other severe heart disease) or accompanying other severe internal diseases (such as uncontrollable diabetes, chronic obstructive pulmonary disease)
7. Patients with prior history of participating in a clinical trial within 30 days from registration for current clinical trial
8. Patient with history of alcohol or drug abuse in the recent 3 months
9. Pregnant women, nursing mothers, or patients of childbearing age who did not agree to contraception (both men and women)
10. Patients with (or suspected to have) abnormality in bile acid secretion (e.g.,. patients with resected gallbladder)
11. Patients who had a history of serious gastrointestinal bleeding, or with diseases that could affect the absorption of oral medication (malabsorption syndrome, active peptic ulcer)
12. Patients with history of severe hypersensitive reaction to active ingredient and excipient of the investigational drug
13. Patient who are in a state that is deemed inappropriate to participate in the clinical trial by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicity(DLT) to determine maximum tolerated dose(MTD) | First cycle of treatment (4-week)
  To determine the dose at which no more than one patient out of up to 6 patients at the same dose level experience a drug-related dose-limiting toxicity

SECONDARY OUTCOMES:
To identify the dose limiting toxicity(DLT) and the safety (toxicity) of DHP107 | First cycle of treatment (4-week)
  Adverse events are evaluated in the first cycle(4-week) according to NCI CTCAE v4.0
To evaluate efficacy(tumor response) by RECIST criteria version 1.1 | every 8 weeks (±1 week)
PK parameters for DHP107 derived from determining their plasma concentrations using validated assays. | First cycle of treatment (4-week)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, M.D., Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryu MH, Ryoo BY, Kim TW, Kim SB, Lim HS, Bae KS, Park SR, Jo YW, Cho HJ, Kang YK. A Phase I/IIa Study of DHP107, a Novel Oral Paclitaxel Formulation, in Patients with Advanced Solid Tumors or Gastric Cancer. Oncologist. 2017 Feb;22(2):129-e8. doi: 10.1634/theoncologist.2016-0273. Epub 2017 Feb 14. PMID 28196905